CLINICAL TRIAL: NCT04483128
Title: Electrical Stimulation With Interferential Current in the Non-especific Chronic Low Back Pain: Effects on the Autonomic Nervous System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Dr. Manuel Albornoz Cabello, Doctor in Physiotherapy (PhD), University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CIFSNA2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Chronic Low-back Pain; Chronic Pain; Autonomic Imbalance
Keywords: electrical stimulation; interferential current; autonomic balance; chronic low back pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with chronic low back pain will be divided into two different groups with 28 patients each:
  * Experimental group: Participants in this group will receive electrical stimulation with interferential current. They will get also instructions to perform core strengthening exercises at home, after variable collection.
  * Control group: Participants in this group will recieve the same electrical stimulation than in the experimental group but with no intensity. This group will get too instructions to perform core strengthening exercises at home (after variable collection) and follow General Practitioner indications about pharmacology.
Who Masked: Participant
Masking Description: Randomization process will be masked by opaques envelopes with numbers. Participants choose one random envelope, unaware the number and group relation. Later, a researcher will associate participants, groups and numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham IFC therapy: Control group (Sham Comparator): This group will recieve also instructions for core strengthening exercises and a single session of interferential current (IFC).
  IFC parameters:
  1. Carrier frequency of 4000 Hz
  2. Amplitude modulated frequency of 65 Hz (AMF)
  3. Sweep frequency of 95 Hz of modulation with a 1:1 swing pattern, in a quadripolar technique.
  4. NO intensity (0 mA)
  5. Session duration: 25 minutes
  Interventions: Device: Electrical stimulation: Interferential Current (IFC): Control Group
- IFC therapy: Experimental group (Experimental): This group will recieve also instructions for core strengthening exercises and a single session of interferential current (IFC).
  IFC parameters:
  1. Carrier frequency of 4000 Hz
  2. Amplitude modulated frequency of 65 Hz (AMF)
  3. Sweep frequency of 95 Hz of modulation with a 1:1 swing pattern, in a quadripolar technique.
  4. Intensity will depend on subjet's tolerance but without generating visible muscle twitches.
  5. Session duration: 25 minutes
  Interventions: Device: Electrical stimulation: Interferential Current (IFC): Experimental Group

INTERVENTIONS:
Device: Electrical stimulation: Interferential Current (IFC): Experimental Group — Application of IFC with Sonopuls 692® (Enraf-Nonius BV, Rotterdam, The Netherlands) device. Parameters:
  1. Carrier frequency of 4000 Hz
  2. Amplitude modulated frequency of 65 Hz (AMF)
  3. Sweep frequency of 95 Hz of modulation with a 1:1 swing pattern, in a quadripolar technique.
  4. Intensity will depend on subjet's tolerance but without generate visible muscle twitches.
  5. Session duration: 25 minutes
  Arms: IFC therapy: Experimental group
Device: Electrical stimulation: Interferential Current (IFC): Control Group — Application of IFC with Sonopuls 692® (Enraf-Nonius BV, Rotterdam, The Netherlands) device. Parameters:
  1. Carrier frequency of 4000 Hz
  2. Amplitude modulated frequency of 65 Hz (AMF)
  3. Sweep frequency of 95 Hz of modulation with a 1:1 swing pattern, in a quadripolar technique.
  4. NO intensity (0 mA)
  5. Session duration: 25 minutes
  Arms: Sham IFC therapy: Control group

SUMMARY:
The aim of this study it's to analyze the relationship between autonomic nervous system balance (ANSb) and chronic pain conditions, especially in this case, non-especific chronic low back pain (CLBP).

Most of physiotherapy approaches focus only in biomechanical aspects, leaving aside what kind of factors could perpetuate CLBP. Since 1985, ANSb was studied due to its potential contribution to chronic pain.

Electrical stimulation, through interferential currents (IFC), it's a safe and well-known therapy used in CLBP with good outcomes regarding pain relief.

The main objective of this study it's to quantify the association between CLBP and ANSb alterations. In second place, the research team aims to record the influence of IFC over pain and ANSb in those subjects.

DETAILED DESCRIPTION:
In the first place, a meeting will be organized with the patients to resolve any doubt about the study and its process. The investigators will make sure every instruction is understandable, giving enough time to read and ask pertinent questions.

Secondly, patients will be provided of an informed consent specific for the present study, according to the legal forms. Participants must agree with all the information and sign the document.

At this point, patients will be interviewed individually by a researcher to collect all the data regarding to the Clinical History in Physiotherapy.

In the next step, patients will be randomized into two different groups by choosing one opaque envelope, containing a number for the allocation. A researcher will make the final allocation depending on the number. Patients were unaware of the group allocation for masking.

This study has to possible groups with a common indication for both:

1. Experimental group: Patients allocated in this group will receive one single session of interferential current (IFC). Current used a carrier frequency of 4.000 Hz, 65Hz of amplitude modulated frequency (AMF) with sweep frecuency of 95Hz in a 1:1 swing pattern (quadripolar technique). Intensity was adjusted according to patient's tolerance without visible muscle twitches. The session will last 25 min.
2. Control group: This group will receive the same intervention than experimental one but with no intensity, for 25 minutes. Patients will keep his general practitioner's indications about pharmacology.
3. Common indication: Both groups will get instructions to perform a set of home-based exercises for core strengthening after variable collecting.

Before and after the session, all the variable measurements will be collected in the same environmental conditions by the same researcher. Basal measurement (before intervention) will be recorded 15 minutes before session for 10 minutes. The second measurement will be taken while the patient recieves the intervention for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with cronic low back pain with at least 3 months of evolution.
* Subjects with a minimal pain of 3/10 according to NPRS
* Subjects with informed consent read and signed.
* Subjects not undergoing any other physical therapy intervention.

Exclusion Criteria:

* Any uncontrolled neurological or cardiac disorder.
* Personal Psychological Apprehension Scale (PPAS) score higher than 37.5.
* Contraindication for electrical stimulation.
* Any regular use of medications known to affect the function of the autonomic nervous system (ANS) or pain perception, including antidepressant, benzodiazepines, anti-inflammatory drugs and beta-blockers, 2 weeks before participating in this study.
* Ineligibility to participate determined by the researches.
* Neurological, musculoskeletal or sensory affectations.
* Evidence of infectious process, fever or hypotension.
* Metallic implants in low back area or treated area
* No surgical interventions in low back area
* Not being under pharmacological treatment with influence in Autonomic Nervous System like antidepressants.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate variability (HRV-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  Heart Rate variability (HRV) is measured by calculating mean HR, maximum HR and minimum HR. First Beat Bodyguard2 device will be used to collect HRV.
Heart Rate variability (HRV-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.
  Heart Rate variability (HRV) is measured by calculating mean HR, maximum HR and minimum HR. First Beat Bodyguard2 device will be used to collect HRV.
Root-mean-square differences of successive heartbeat intervals (RMSSD-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  RMSSD it's an indirect indicator of parasympathic nervous system level of activity. First Beat Bodyguard2 device will be used to collect RMSSD.
Root-mean-square differences of successive heartbeat intervals (RMSSD-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.
  RMSSD it's an indirect indicator of parasympathic nervous system level of activity. First Beat Bodyguard2 device will be used to collect RMSSD.
Standard Deviation 1 (SD1-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  SD1 is an indicator of the autonomic nervous balance. First Beat Bodyguard2 device will be used to collect it.
Standard Deviation 1 (SD1-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.
  SD1 is an indicator of the autonomic nervous balance. First Beat Bodyguard2 device will be used to collect it.
Standard Deviation 2 (SD2-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  SD2 is an indicator of the autonomic nervous balance. First Beat Bodyguard2 device will be used to collect it.
Standard Deviation 2 (SD2-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.s.
  SD2 is an indicator of the autonomic nervous balance. First Beat Bodyguard2 device will be used to collect it.
Stress Index (SS-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  SS it's an indicator of sympathetic nervous system level of activation. First Beat Bodyguard2 device will be used to collect SS.
Stress Index (SS-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.s.
  SS it's an indicator of sympathetic nervous system level of activation. First Beat Bodyguard2 device will be used to collect SS.
Sympathetic / Parasympathetic Ratio (S/PS Ratio-a) | Evaluation before intervention (basal): 15 minutes before intervention, for 10 minutes.
  S/PS Ratio it's an indicator of autonomic nervous system balance. First Beat Bodyguard2 device will be used to collect S/PS Ratio.
Sympathetic / Parasympathetic Ratio (S/PS Ratio-b) | Evaluation during the intervention: For 20 minutes, while the interferential current (intervention) is being applied.s.
  S/PS Ratio it's an indicator of autonomic nervous system balance. First Beat Bodyguard2 device will be used to collect S/PS Ratio.
Numeric Pain Rating Scale (NPRS-a) | Evaluation before intervention (basal): 15 minutes before intervention.
  NPRS it's an scale used to measure with ease, patient's perceived pain with a scoring of 0 (no pain) and 10 (maximum pain).
Numeric Pain Rating Scale (NPRS-b) | Evaluation immediately after treatment session.
  NPRS it's an scale used to measure with ease, patient's perceived pain with a scoring of 0 (no pain) and 10 (maximum pain).

SECONDARY OUTCOMES:
Roland Morris Questionnaire (RMQ-a) | Evaluation before intervention (basal): 15 minutes before intervention.
  RMQ it's a questionnaire used to measure an individual level of disability related to low back pain, with a scoring of 0 (no disability at all) and 24 (maximum disability).
Roland Morris Questionnaire (RMQ-b) | Evaluation immediately after treatment session.
  RMQ it's a questionnaire used to measure an individual level of disability related to low back pain, with a scoring of 0 (no disability at all) and 24 (maximum disability).
Scale for Personal Psychological Apprehension (SPPA) | Evaluation before intervention (basal): 15 minutes before intervention.
  SPPA it's a questionnaire made to measure subject's susceptibility to receive electrical stimulation. A scoring of >45 points indicates that subject shouldnt be treated with electrical therapy.
Dosimetry achieved with electrical stimulation | Recorded immediately after treatment session.
  Maximal dosimetry reached during the session will be recorded in mA.

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Albornoz Cabello, Seville, Spain

IPD SHARING:
Plan to Share IPD: No